CLINICAL TRIAL: NCT06910566
Title: A Prospective Study on the Factors Sustaining Tobacco Abstinence in Patients Treated With Radio-chemotherapy or Radiotherapy Alone for Head and Neck or Lung Cancer
Brief Title: Factors Sustaining Tobacco Abstinence in Cancer Patients Treated With Radio-chemotherapy or Radiotherapy
Acronym: TABAC STOP ORL
Status: Recruiting | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: TABAC STOP ORL POUMON-20-001; 2020-A02912-37 (Other: ANSM)
Record Dates: First submitted 2025-03-19; First posted 2025-04-04 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-03

CONDITIONS: Smoking Cessation; Nicotine Addiction; Nicotine Dependence; Smoking; Head and Neck Neoplasms
Keywords: Tobacco abstinence; Head and neck cancer; Smoking cessation; Nicotine dependence; Cancer treatment
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Smoking; Head and Neck Neoplasms | interventions — Chemoradiotherapy; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Chemoradiotherapy or radiotherapy alone — Patients included in the study receive standard treatment with chemoradiotherapy or radiotherapy alone for their head and neck cancer or lung cancer. These treatments are part of their routine care and are not part of the observational study.
  Other Names: chemoradiotherapy; radiotherapy

SUMMARY:
The TABAC STOP ORL POUMON study aims to evaluate the factors influencing long-term smoking cessation in patients with head and neck cancer (HNC) or lung cancer undergoing radiotherapy or chemoradiotherapy. This is a single-center observational study, following patients at 1, 6, and 12 months after treatment completion. The primary objective is to determine the proportion of abstinent patients at 6 months, while secondary objectives analyze factors influencing abstinence, smoking trajectories, and reasons for relapse. A total of 100 patients will be included to ensure robust statistical analysis.

DETAILED DESCRIPTION:
The TABAC STOP ORL POUMON study is a prospective, single-center observational study aiming to understand factors influencing long-term smoking cessation in patients treated for head and neck or lung cancer. Tobacco is a leading cause of death and disease, particularly in areas like Hauts-de-France with high smoking rates.

Eligible patients, undergoing radiotherapy or chemoradiotherapy, are enrolled during the final week of treatment, completing questionnaires assessing nicotine dependence and alcohol use. Follow-ups are scheduled at 1, 6, and 12 months, through clinic visits or phone interviews.

The primary endpoint is the proportion of patients who remain smoke-free at 6 months. Secondary endpoints include factors influencing smoking cessation, reasons for relapse, and changes in nicotine and alcohol dependence. The study will enroll 100 patients, expecting 81 evaluable cases, with data quality ensured through regular checks and source verification.

ELIGIBILITY:
Inclusion Criteria :

* Patient aged 18 years or older
* Diagnosed with head and neck cancer or lung cancer
* Undergoing curative treatment with chemoradiotherapy, radiotherapy alone, or stereotactic radiotherapy
* Current or former smoker
* Patient covered by a social security scheme
* Patient informed and having given consent for data collection

Patients with human papillomavirus (HPV) may also be included

Exclusion Criteria :

* Patient receiving palliative treatment
* Patient under guardianship or curatorship

Study Exit Criteria :

- Protocol-defined exit : After the 12-month consultation

Early exit :

* Withdrawal of consent for data collection
* Death of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients diagnosed with head and neck cancer (HNC) or lung cancer, who are undergoing curative treatment with chemoradiotherapy, radiotherapy alone, or stereotactic radiotherapy at the Centre Oscar Lambret in Lille, France. Participants are current or former smokers and are recruited during the last week of their radiotherapy treatment. The study aims to evaluate factors associated with maintaining tobacco abstinence in this specific patient population, focusing on their smoking cessation journey following cancer treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Abstinence at 1 month and 6 months after the end of treatment | 1 and 6 months after the end of treatment.
  The primary outcome measure will be abstinence at 1 month (physical consultation or telephone follow-up) and at 6 months after the end of treatment.

SECONDARY OUTCOMES:
Proportion of patients willing to attend a smoking cessation consultation | At the 1-month telephone follow-up after the end of treatment.
  Evaluation of patients willing to attend a smoking cessation consultation (assessed among active smokers at the phone follow-up consultation).
Abstinence at 1 month after the end of treatment | 1 month after the end of treatment
  Proportion of tobacco-abstinent patients 1 month after the end of radiotherapy or chemoradiotherapy
Abstinence at 6 months after the end of treatment | 6 months after the end of treatment
  Proportion of tobacco-abstinent patients 6 months after the end of radiotherapy or chemoradiotherapy
Abstinence at 12 months after the end of treatment | 12 months after the end of treatment
  Proportion of tobacco-abstinent patients 12 months after the end of radiotherapy or chemoradiotherapy
Cigarette dependence (Cigarette Dependence Scale, CDS) | Baseline
  Level of nicotine dependence assessed using the Cigarette Dependence Scale (CDS). The CDS is a validated 12-item scale with scores ranging from 0 to 60, where higher scores indicate dependence.
Alcohol use and dependence (Alcohol Use Disorders Identification Test, AUDIT) | Baseline
  Alcohol consumption and dependence assessed using the Alcohol Use Disorders Identification Test (AUDIT). The AUDIT is a 10-item scale with scores ranging from 0 to 40, where higher scores indicate higher risk of alcohol-related harm.

CONTACTS AND LOCATIONS:
Overall Officials: Gautier LEFEBVRE, MD, Study Director — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No